CLINICAL TRIAL: NCT07327177
Title: The Effects of Blood Flow Restriction Rope Training on Athletic Performance, Muscle Strength, and Hypertrophy in Male Volleyball Players
Brief Title: BFR Rope Training in Male Volleyball Players
Acronym: 8wBFR_rope
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Neslihan AKÇAY, Assoc. Prof. Dr., Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKarabuk-5
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Volleyball; Performance; Power
Keywords: blood flow restriction; rope; volleyball; hypertrophy
MeSH Terms: conditions — Hypertrophy | interventions — Blood Pressure; Muscle Strength; Blood Flow Restriction Therapy; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor) Participants were strictly separated and think their intervention is the main intervention. The same is true for care providers. Outcome assessors were unaware of participant group status and were not allowed to ask correspondingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- Blood Pressure (Other): Determination of Blood Pressure
  Interventions: Other: Blood Pressure
- Muscle Strength (Experimental): Determination of Muscle Strength
  Interventions: Other: Muscle Strength
- Serve Speed (Other): Determination of Serve Speed
  Interventions: Other: Serve Speed
- Blood Flow Restriction (BFR) (Other): Blood Flow Restriction Protocol
  Interventions: Other: Blood Flow Restriction
- Rating of Perceived Exertion (RPE) (Other): Determination of Perceived Exertion
  Interventions: Other: Rating of Perceived Exertion
- Battle Rope Training (Other): Battle Rope Training Protocol
  Interventions: Other: Battle Rope Training
- Arm Circumference (Other): Arm Circumference Measurement
  Interventions: Other: Arm Circumference
- Skeletal Muscle Endurance (Other): Skeletal Muscle Endurance Tests (Sit-Up, Push-Up, and Pull-Up)
  Interventions: Other: Skeletal Muscle Endurance
- Anaerobic Power (Other): Anaerobic Power Assessment
  Interventions: Other: Anaerobic Power
- Bench Press 1RM Test (Other): Bench Press 1RM Test Measurement
  Interventions: Other: Bench Press 1RM Test
- Triceps Push-Down 1RM Test (Other): Triceps Push-Down 1RM Test Measurement
  Interventions: Other: Triceps Push-Down 1RM Test
- Hand Grip Strength Test (Other): Hand Grip Strength Test Measurement
  Interventions: Other: Hand Grip Strength Test
- Yo-Yo IR1 Test (Other): Yo-Yo IR1 Test Measurement
  Interventions: Other: Yo-Yo IR1 Test
- Ultrasound (US) (Other): Ultrasound (US) Measurements
  Interventions: Other: Ultrasound (US)
- Perceived Discomfort Level (Other): Determination of Perceived Discomfort Level
  Interventions: Other: Perceived Discomfort Level
- Exercise Enjoyment (Other): Exercise Enjoyment Assessment
  Interventions: Other: Exercise Enjoyment
- Perceived Exertion Level (OMNI-RES) (Other): Perceived Exertion Level Assessment
  Interventions: Other: Perceived Exertion Level (OMNI-RES)

INTERVENTIONS:
Other: Blood Pressure — A digital Omron device (model M2; Ankara, Turkey) will be used to measure participants' resting blood pressure. Prior to exercise, systolic, diastolic, and heart rate values will be recorded, and individuals outside the 140/90 mmHg range will be excluded. Participants will remain seated for 10 minutes, after which three measurements will be taken from the dominant arm with at least 1 minute between readings. Resting blood pressure will be calculated as the average of these three values, following American Heart Association guidelines (Pickering et al., 2005).
  Arms: Blood Pressure
Other: Muscle Strength — Dominant and non-dominant shoulder internal and external rotation strength will be assessed using a Lafayette digital handheld dynamometer. This portable device provides peak force, time to peak force, total test duration, and average force in kilograms, Newtons, and pounds. Participants will receive verbal instructions and complete a familiarization trial before testing. The "make test" technique will be used, in which the examiner stabilizes the device while the participant applies maximal isometric force. All measurements will be taken twice by the same trainer. Prior to testing, a 10-minute warm-up including upper-extremity and shoulder rotation movements will be performed. Participants will then lie supine on a flat surface, and dominant and non-dominant internal and external rotation strength will be measured and recorded (Kesilmiş & Manolya, 2020).
  Arms: Muscle Strength
Other: Serve Speed — The serve speed test will be conducted in the Hasan Doğan Sports Sciences Gymnasium at Karabük University using official balls (FIVB Beach Championship VLS300 MIKASA). Athletes will begin with a 15-minute warm-up consisting of joint mobility exercises (e.g., knee flexion/extension, shoulder rotation, ankle dorsiflexion), followed by technical movements such as ball-free jumping and running to enhance coordination. Each player will then perform ten practice serves. A total of 196 power-kick serves (28 per participant) will be recorded without opposition. After each isometric exercise, participants will execute four maximal-intensity serves, and ball speed will be determined from these attempts. Athletes will be encouraged to strike the ball with maximum force. A radar device will be positioned 8 m behind the service line and 3 m above the ground to capture serve velocity at a height consistent with ball-hand contact (Buscà et al., 2012). Serve speed will be measured using a standard ra
  Arms: Serve Speed
Other: Blood Flow Restriction — The arterial occlusion pressures (AOP) of the athletes randomized to the experimental group will be automatically determined using a digital LED-display BFR device (Fit Cuffs BFR, Denmark). Optimal cuff width, occlusion pressure, and exercise procedures have been previously described in the literature (Loenneke et al., 2015; Scott et al., 2015). A 4-inch-wide tourniquet will be applied to the upper arm of the participant's dominant limb. During the exercise, the AOP will be maintained at 60% using the Fit Cuffs BFR Unit (Denmark), and consistent pressure will be applied to the limb throughout the full range of motion. All participants will use the same cuff model, and 60% AOP will be administered with an FDA/CE-approved automatic Smart Cuffs Pro device (Elite, USA), applied to the proximal region of the arm.
  Arms: Blood Flow Restriction (BFR)
Other: Rating of Perceived Exertion — After each training session, RPE will be collected using the 6-20 Borg Scale at the end of the session, where 6 indicates "no exertion" and 20 indicates "maximal exertion" (Foster et al., 2021).
  Arms: Rating of Perceived Exertion (RPE)
Other: Battle Rope Training — Based on prior literature recommending battle ropes measuring 12-15 m in length, 3-5 cm in diameter, and 9-16 kg in weight (Pustina et al., 2017; Tessitore et al., 2006; Ziy et al., 2009), this study will use a 12-m, 3.8-cm diameter, 12-kg rope. Participants will perform wave-style rope exercises in a standing position with feet shoulder-width apart and the trunk flexed forward at approximately 30-45°. The rope will be anchored at its midpoint to a stable object, and participants will grip the ends (5 m ± 5 cm each) and execute bilateral oscillations. The protocol will include three sets of five exercises, with progressive durations across the 8-week period: 15 seconds in Weeks 1-2, 20 seconds in Weeks 3-5, and 25 seconds in Weeks 6-8. Rest intervals between sets will remain consistent at 45 seconds throughout the training program.
  Arms: Battle Rope Training
Other: Arm Circumference — Before the training session and without performing any physical activity, arm circumference will be measured using a 300-cm non-elastic measuring tape. Measurements will be taken at a 90° elbow angle from the midpoint of the upper arm, over the biceps muscle (Otman, 2003).
  Arms: Arm Circumference
Other: Skeletal Muscle Endurance — Upper-body and trunk muscular endurance will be assessed using standardized ACSM protocols. Upper-body endurance will be measured with the ACSM push-up test: men will perform standard push-ups, while women will complete kneeling push-ups. The test will stop at volitional fatigue or after two consecutive form errors (chin to mat and full elbow extension). Trunk endurance will be evaluated using the cadence-based YMCA bent-knee sit-up test, performed at one repetition every 2 seconds until volitional fatigue. A valid sit-up requires elbows touching the knees and returning to the starting position in cadence. Upper-body pulling endurance will be tested with a pronated-grip pull-up test. Repetitions must include the chin rising above the bar and full controlled elbow extension. The test ends at volitional fatigue or after repeated form errors. All endurance tests (push-up, sit-up, pull-up) will be performed to volitional fatigue with 2-3 minutes of rest between tests, and the same test
  Arms: Skeletal Muscle Endurance
Other: Anaerobic Power — The Wingate Anaerobic Power Test (WAnT) is a widely used 30-second cycling test designed to measure short-term, high-intensity power output and anaerobic energy system capacity (Reiser et al., 2002). Conducted on a Monark 894E ergometer, the test uses a resistance load adjusted to each participant's body mass (Jaafar et al., 2014). Before testing, participants will complete a 4-5 minute warm-up at 60-70 W and 60-70 rpm, including 2-3 short sprints, followed by 3-5 minutes of passive rest. Saddle and handlebar settings will be adjusted so the knee reaches full extension at the lowest pedal position, and feet will be secured with clips. Participants will accelerate to maximal speed without resistance; once they reach 150 rpm, the programmed resistance load will automatically engage. They will then pedal maximally for 30 seconds against this resistance while receiving verbal encouragement (Ozkan, 2007).
  Arms: Anaerobic Power
Other: Bench Press 1RM Test — Participants will begin with a 5-minute treadmill warm-up at 9 km/h followed by three minutes of light stretching (do Carmo et al., 2021). A specific warm-up will then be performed: 5 reps at 50% of estimated 1RM, followed by 1-2 sets of 2-3 reps at 60-80%. After warm-up, participants will perform single-rep attempts with gradually increasing loads to determine their 1RM, resting 3-5 minutes between trials. Up to five attempts will be used to identify the true 1RM (Schoenfeld et al., 2016).
  Arms: Bench Press 1RM Test
Other: Triceps Push-Down 1RM Test — Participants will stand in front of the triceps push-down machine, gripping the bar with a shoulder-width pronated grip. Throughout the exercise, the arms will be kept close to the torso, with the trunk slightly leaned forward, ensuring that the hands do not touch the body during full elbow extension. Participants will push the bar downward until reaching full elbow extension, then return to the starting position in a controlled manner; this will count as one repetition. The maximum load that each participant can successfully lift for one full repetition will be recorded as their 1RM (Hussain et al., 2020).
  Arms: Triceps Push-Down 1RM Test
Other: Hand Grip Strength Test — A calibrated hand grip dynamometer (Takei 5101, Tokyo, Japan) will be used to evaluate maximal hand grip strength. Participants will be instructed to grasp the dynamometer with their hand while exerting maximal isometric force, maintaining extended elbows and a neutral wrist position at the lateral side of the body. The testing protocol will include two trials with a 60-second rest interval between them. The highest value obtained will be recorded as the maximal force output. Throughout the test, participants will be strongly encouraged to exert maximal effort (Lopes-Silva et al., 2022).
  Arms: Hand Grip Strength Test
Other: Yo-Yo IR1 Test — The Yo-Yo Intermittent Recovery Level 1 (Yo-Yo IR1) test will be used to assess intermittent endurance capacity (Krustrup et al., 2003). Participants will complete 20 m shuttle runs at progressively increasing speeds, with 10 seconds of active recovery (light jogging over 2 m × 5 m) between runs. The test will stop when the participant can no longer maintain the required pace or fails to reach the line on time for two consecutive shuttles. Performance will be scored by the total distance (number of completed shuttles). A familiarization trial will be conducted before testing. The Yo-Yo IR1 demonstrates high reliability (ICC = 0.94; CV = 3.6%) (Krustrup et al., 2003).
  Arms: Yo-Yo IR1 Test
Other: Ultrasound (US) — Muscle thickness and cross-sectional area (CSA) will be measured 48-72 hours after the final training session, with no prior physical activity. A blinded physician will conduct all assessments using standardized anatomical points for the biceps brachii, triceps brachii, brachialis, anterior deltoid, upper trapezius, and rectus abdominis. Measurements will be taken in the axial plane with a light, 90° probe contact. A Toshiba Aplio 500 ultrasound device (10 MHz linear probe) will be used. CSA will be calculated by tracing the inner muscle border, and muscle thickness will be measured between superficial and deep aponeuroses. Two radiology specialists will evaluate the results jointly (Kubo et al., 2011).
  Arms: Ultrasound (US)
Other: Perceived Discomfort Level — Perceived Discomfort Level (PDL) will be assessed using a scale ranging from 0 ("no discomfort") to 10 ("maximum discomfort") (Borg, 1998). The PDL will be evaluated twice: once for overall body discomfort and once specifically for arm discomfort.
  Arms: Perceived Discomfort Level
Other: Exercise Enjoyment — Exercise enjoyment will be measured using the shortened 8-item version of the Physical Activity Enjoyment Scale (PACES), originally developed by Kendzierski and DeCarlo (1991) and later adapted by Raedeke (2007). This single-factor scale evaluates the level of enjoyment experienced during exercise. Each item is rated on a 7-point Likert scale ranging from 1 ("do not enjoy at all") to 7 ("enjoy very much"), with 4 representing a neutral midpoint. Higher scores indicate greater enjoyment derived from the physical activity (Soylu et al., 2023).
  Arms: Exercise Enjoyment
Other: Perceived Exertion Level (OMNI-RES) — The OMNI-RES resistance exercise scale will be used to assess participants' perceived exertion levels. A rating will be recorded at the end of each set, and the average of all set scores will be calculated and documented at the end of the exercise session. The scale will remain within the participant's visual field throughout the session, and they will be instructed to focus on their sense of effort immediately before each rating. Using standardized definitions and instructions, participants will rate their exertion on a scale ranging from 0 ("extremely easy") to 10 ("extremely hard") (Robertson et al., 2003).
  Arms: Perceived Exertion Level (OMNI-RES)

SUMMARY:
The study will be conducted during the preparatory period of the volleyball players and will span eight weeks. Throughout this period, athletes will continue their regular volleyball training four days per week, while the experimental group (n = 10) will perform rope training with blood flow restriction (BFR) twice per week, and the control group (n = 10) will perform the same rope training without BFR. Assessments will be carried out at the beginning of the 8-week period (pre-test) and at the end of the intervention (post-test). For both groups, all exercises will target the upper-extremity muscle groups. During the study, participants will be instructed to avoid consuming any medications, engaging in additional strenuous physical activities, and using any techniques or ergogenic aids that might influence the results. In both testing sessions, a standardized warm-up protocol will be implemented, consisting of a 5-minute treadmill run at 9 km/h on a Sprint Runner device (Hoggan Health Industries, Draper, UT), followed by 3 minutes of light full-body stretching. This warm-up procedure will be applied consistently across both groups to ensure standardization.

DETAILED DESCRIPTION:
This study aims to investigate the effects of blood flow restriction (BFR) rope training on athletic performance, muscle strength, and muscle hypertrophy in male volleyball players through an eight-week intervention. Conducted during the athletes' preparatory period, the study requires participants to perform rope-training sessions four days per week in addition to their regular volleyball training. On the first day, all athletes will undergo anthropometric measurements, and a familiarization session will be conducted to minimize potential learning effects. Participants will then be randomly assigned to either a BFR rope-training experimental group (BFR) or a control group (CON) performing standard rope training. Both groups will follow a progressive training protocol consisting of three sets and five exercises, while the BFR group will train under a cuff pressure set at 60% of limb occlusion pressure (LOP). Throughout the training sessions, heart rate, rating of perceived exertion (RPE), perceived discomfort (PD), OMNI-RES exercise difficulty, and PACES exercise enjoyment scores will be recorded. Pre- and post-intervention assessments will include ultrasound measurements of muscle thickness and cross-sectional area, one-repetition maximum (1RM) tests for biceps and triceps, upper-body strength tests (push-ups, sit-ups, and squats), shoulder strength using a Lafayette device, handgrip strength, aerobic endurance via the Yo-Yo IR1 test, anaerobic performance via the Wingate test, and volleyball serve speed measurements. All exercises will target upper-extremity muscle groups, and participants will be instructed to refrain from using any medications, ergogenic aids, or additional strenuous exercise that could influence outcomes. During both pre- and post-testing sessions, all athletes will complete a standardized warm-up protocol consisting of a 5-minute treadmill run at 9 km/h followed by 3 minutes of light full-body stretching. This comprehensive design aims to provide valuable insights into how BFR-based rope training influences performance adaptations in volleyball athletes.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Male volleyball athletes
* Willing to maintain the intervention for all sessions

Exclusion Criteria:

* Being under 18 years old
* Having a chronic disease
* Contraindications for exercise

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Muscle Thickness (Ultrasound) - Biceps, Triceps, Brachialis, Antrerior Deltoid, Upper Trapezius, Rectus Abdominis | From baseline assessment to 8-week follow-up assessment
  Change in muscle thickness (mm) from baseline to 8-week follow-up as measured by diagnostic ultrasound.
Muscle Cross-Sectional Area (CSA) - Biceps, Triceps, Brachialis, Antrerior Deltoid, Upper Trapezius, Rectus Abdominis | From baseline assessment to 8-week follow-up assessment.
  Change in muscle CSA (cm²) for specified muscles combined or reported individually from baseline to 8-week follow-up as measured by diagnostic ultrasound.
1-Repetition Maximum (1RM) - Bench Press and Triceps Push-Down | From baseline assessment to 8-week follow-up assessment.
  Change in bench Press and triceps push-down 1RM (kg) from baseline to 8-week follow-up.
Shoulder Internal/External Rotation Strength | From baseline assessment to 8-week follow-up assessment
  Change in peak isometric rotation force (kg) for dominant and non-dominant shoulders (measured by handheld dynamometer, make test) from baseline to 8-week follow-up.
Hand Grip Strength | From baseline assessment to 8-week follow-up assessment.
  Change in maximal handgrip strength (kg) from baseline to 8-week follow-up measured with a calibrated dynamometer
Upper-Body Muscular Endurance - Push-Up, Sit-Up, Pull-Up | From baseline assessment to 8-week follow-up assessment
  Change in number of repetitions to volitional fatigue for push-up, sit-up, and pull-up tests from baseline to 8-week follow-up.
Serve Speed | From baseline assessment to 8-week follow-up assessment
  Change in maximum volleyball serve speed (km/h) from baseline to 8-week follow-up measured by radar.
Aerobic Intermittent Endurance - Yo-Yo IR1 | From baseline assessment to 8-week follow-up assessment
  Change in Yo-Yo IR1 performance (VO2max) from baseline to 8-week follow-up.
Anaerobic Power - Wingate Test | From baseline assessment to 8-week follow-up assessment
  Change in peak power and mean power (W and W·kg-¹) derived from the 30-s Wingate test from baseline to 8-week follow-up.
Perceived Exertion - RPE (Borg 6-20) | From baseline assessment to 8-week follow-up assessment
  Change in session RPE (Borg 6-20 score), averaged across training sessions, from baseline to 8-week follow-up.
Perceived Discomfort (RPD) | From baseline assessment to 8-week follow-up assessment
  Change in perceived discomfort scores (0-10 scale) for whole body and arm-specific measures from baseline to 8-week follow-up.
Exercise Enjoyment (PACES) | From baseline assessment to 8-week follow-up assessment
  Change in exercise enjoyment score (8-item PACES, score range 1-7) from baseline to 8-week follow-up.
OMNI-RES (Resistance Exercise Perceived Exertion) | From baseline assessment to 8-week follow-up assessment
  Change in OMNI-RES average score (0-10) across sessions from baseline to 8-week follow-up.

SECONDARY OUTCOMES:
Anthropometric Measurements 1 | Baseline
  Participants' height (cm) will assess by using a stadiometer (Holtain Stadiometer, England).
Anthropometric Measurements 2 | Baseline
  Body weight (kg) will asses by Inbody 270 (Biospace, California, USA)
Anthropometric Measurements 3 | Baseline
  Body mass index (BMI) (kg/m2) will asses by Inbody 270 (Biospace, California, USA).
Anthropometric Measurements 4 | Baseline
  Body fat percentage (%) will asses by Inbody 270 (Biospace, California, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Akçay, Doctorate, Study Chair — Karabuk University
Locations (1):
- Karabuk University, Karabük, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kamis O, Rolnick N, de Queiros VS, Akcay N, Keskin K, Yildiz KC, Sofuoglu C, Werner T, Hughes L. Impact of limb occlusion pressure assessment position on performance, cardiovascular, and perceptual responses in blood flow restricted low-load resistance exercise: A randomized crossover trial. J Sports Sci. 2025 Oct;43(19):2256-2264. doi: 10.1080/02640414.2024.2422205. Epub 2024 Nov 10. PMID 39523480
- [Result] Keskin K, Akcay N, Ozmen T, Contarli N, Yildiz KC, Sofuoglu C, Kamis O, Rolnick N, de Queiros VS, Montoye A. Effects of different pre-exercise strategies on jumping performance in female volleyball players. J Sports Med Phys Fitness. 2025 Jan;65(1):59-68. doi: 10.23736/S0022-4707.24.16196-8. Epub 2024 Oct 3. PMID 39360986